CLINICAL TRIAL: NCT04361760
Title: Better to Focus or to Spread? Signal Propagation and Its Relationship to Cognitive Performance in the Aging Human Brain
Brief Title: Signal Propagation and Its Relationship to Cognitive Performance in the Aging Human Brain (Focus or Spread)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: 2020-00258
Record Dates: First submitted 2020-04-22; First posted 2020-04-24 (Actual); Last update posted 2021-10-05 (Actual); Status verified 2021-10

CONDITIONS: Healthy Aging
Keywords: transcranial magnetic stimulation (TMS); high-density electroencephalography (hd-EEG); simultaneous TMS-hd-EEG; diffusion tensor imaging (DTI); neural dedifferentiation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Healthy younger participants (20-30y) (Experimental): Within-subject design. In a visual discrimination task participants will be asked to identify specific features of visual stimuli (i.e., the gender of a face, or the motion direction of a grating). During this task, single-pulse TMS will be applied in one-third of the trials; sham stimulation will be applied in a further third of the trials; and no stimulation will be applied in the remaining third of the trials, while hd-EEG will be continuously measured. The order of these three stimulation conditions (i.e., single-pulse TMS, sham, or no stimulation, during the 1st, 2nd, or 3rd third of the trials) will be counterbalanced over participants.
  Interventions: Device: single-puls TMS; Device: sham stimulation
- Healthy older participants (65-75y) (Experimental): Within-subject design. In a visual discrimination task participants will be asked to identify specific features of visual stimuli (i.e., the gender of a face, or the motion direction of a grating). During this task, single-pulse TMS will be applied in one-third of the trials; sham stimulation will be applied in a further third of the trials; and no stimulation will be applied in the remaining third of the trials, while hd-EEG will be continuously measured. The order of these three stimulation conditions (i.e., single-pulse TMS, sham, or no stimulation, during the 1st, 2nd, or 3rd third of the trials) will be counterbalanced over participants.
  Interventions: Device: single-puls TMS; Device: sham stimulation

INTERVENTIONS:
Device: single-puls TMS — Medical Device (MD): MagPro X100
Device: sham stimulation — Sham stimulation is delivered with a dedicated coil, which is magnetically shielded and thus produces only approx. 20% of the nominal magnetic field. This is not enough to reach and stimulate the cortex, but the produced sound and scalp sensation are the same as with a real TMS coil.

SUMMARY:
In the next three decades, the world's population over 60 years old is expected to more than double its size. Even in the absence of an obvious pathology (i.e., healthy aging), advancing age is typically associated with a progressive decline in cognitive performance. Although pathophysiological changes in age-related neurodegenerative disorders have received much attention over the past years, far less is known about the neural processes affecting cognition in healthy ageing. One of these postulated processes is neural dedifferentiation (i.e., a decrease in neural selectivity, by which neural representations of processed information become less univocally distinguishable), possibly accompanied by the recruitment of additional cortical areas in the healthy aging brain. To date, these processes have been extensively studied on the neural level, yet their functional significance for cognitive behaviour remains largely unclear. This project will investigate neural dedifferentiation and its relationship to cognitive performance in the healthy aging brain. To this end, the investigators will use a combination of state-of-the-art technologies including simultaneous transcranial magnetic stimulation (TMS) and high-density electroencephalography (hd-EEG) as well as diffusion tensor imaging (DTI). Perspectives include a better understanding of the relationship between neurophysiological mechanisms and cognitive performance in the healthy aging brain.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent as documented by signature
* Age between 20-30 or 65-75 years
* Neurologically healthy, i.e., with no documented or present neurological disease or brain injury
* Normal or corrected-to-normal visual acuity

Exclusion Criteria:

* Any instable medical condition, in particular epilepsy (past or present, including seizures or febrile convulsions)
* Any surgical intervention to the brain
* Heart diseases
* Implanted medical devices (e.g., cochlear implants, infusion pumps, neurostimulators, pacemakers)
* History of migraine or strong headaches
* Sleep deprivation
* Presence of non-MRI safe metal in the body
* Drug or alcohol abuse
* Intake of any medication that is likely to lower seizure threshold
* Claustrophobia
* For female participants: in order to participate in the study, female participants in reproductive age need to take a pregnancy test (a standard urine pregnancy test will be provided).
* For female participants: breastfeeding
* Inability to follow the procedures of the study, e.g. due to language problems, psychological disorders, etc. of the participant
* Lack of knowledge of the German language
* Participation in another study with investigational drug within the 30 days preceding and during the present study
* Previous enrolment into the current study
* Enrolment of the investigator, his/her family members, employees and other dependent persons

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2020-06-25 (Actual); Primary Completion 2021-04-08 (Actual); Study Completion 2021-05-18 (Actual)

PRIMARY OUTCOMES:
Age-related differences in the spatio-temporal patterns of signal propagation | 2 hours
  The spatiotemporal patterns of signal propagation, as measured with a combined TMS-hd-EEG approach, in younger and older healthy participants, reflecting age-related differences on the neural level.

SECONDARY OUTCOMES:
Association between the performance in a cognitive test battery and patterns of signal propagation in younger and older participants | 4 hours
  The association between the performance in a specific cognitive test and the aforementioned patterns of signal propagation in younger and older healthy participants, reflecting the functional significance of these age-related patterns on the cognitive level.
Association between the performance in a cognitive test battery and patterns of signal propagation in better- and worse-performers | 4 hours
  The association between the performance in a specific cognitive test and the aforementioned patterns of signal propagation in better- and worse-performers, reflecting the functional significance of these age-independent patterns on the cognitive level.
Association between the patterns of signal propagation and the structural properties of the white matter | 4 hours
  The association between the aforementioned patterns of signal propagation and the structural properties of the white matter interconnecting the involved cortical areas, as measured by DTI.

CONTACTS AND LOCATIONS:
Overall Officials: René M. Müri, Prof. Dr., Principal Investigator — Department of Neurology, Inselspital, Bern University Hospital
Locations (1):
- Department of Neurology, Inselspital, Bern University Hospital, Bern, Switzerland

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Background] Hedden T, Gabrieli JD. Insights into the ageing mind: a view from cognitive neuroscience. Nat Rev Neurosci. 2004 Feb;5(2):87-96. doi: 10.1038/nrn1323. No abstract available. PMID 14735112
- [Background] Raz N, Rodrigue KM. Differential aging of the brain: patterns, cognitive correlates and modifiers. Neurosci Biobehav Rev. 2006;30(6):730-48. doi: 10.1016/j.neubiorev.2006.07.001. Epub 2006 Aug 17. PMID 16919333
- [Background] Park J, Carp J, Kennedy KM, Rodrigue KM, Bischof GN, Huang CM, Rieck JR, Polk TA, Park DC. Neural broadening or neural attenuation? Investigating age-related dedifferentiation in the face network in a large lifespan sample. J Neurosci. 2012 Feb 8;32(6):2154-8. doi: 10.1523/JNEUROSCI.4494-11.2012. PMID 22323727
- [Background] Sala-Llonch R, Bartres-Faz D, Junque C. Reorganization of brain networks in aging: a review of functional connectivity studies. Front Psychol. 2015 May 21;6:663. doi: 10.3389/fpsyg.2015.00663. eCollection 2015. PMID 26052298
- [Background] Ziemann U. Transcranial magnetic stimulation at the interface with other techniques: a powerful tool for studying the human cortex. Neuroscientist. 2011 Aug;17(4):368-81. doi: 10.1177/1073858410390225. Epub 2011 Feb 10. PMID 21311054
- [Background] Ozdemir RA, Tadayon E, Boucher P, Momi D, Karakhanyan KA, Fox MD, Halko MA, Pascual-Leone A, Shafi MM, Santarnecchi E. Individualized perturbation of the human connectome reveals reproducible biomarkers of network dynamics relevant to cognition. Proc Natl Acad Sci U S A. 2020 Apr 7;117(14):8115-8125. doi: 10.1073/pnas.1911240117. Epub 2020 Mar 19. PMID 32193345